CLINICAL TRIAL: NCT03862716
Title: Remission Evaluation of a Metabolic Intervention for Type 2 Diabetes With IDegLira (REMIT IDegLira): A Randomized Controlled Trial
Brief Title: Remission Evaluation of a Metabolic Intervention for Type 2 Diabetes With IDegLira
Acronym: REMITiDegLira
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMITiDegLira
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; IDegLira; Metformin; Insulin; Diet; Excercise; Lifestyle
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — IDegLira; insulin degludec; Metformin; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Drug: IDegLira - sc injection; Drug: metformin - oral administration; Drug: insulin degludec - sc injection; Behavioral: lifestyle therapy, diet and exercise
  Interventions: Drug: IDegLira; Drug: insulin degludec; Drug: Metformin; Behavioral: Lifestyle Therapy
- Standard Care (No Intervention): Standard glycemic care as informed by the current clinical practice guidelines

INTERVENTIONS:
Drug: IDegLira — Dose is titrated to achieve fasting normoglycemia
  Other Names: insulin degludec / liraglutide
  Arms: Intervention
Drug: insulin degludec — In those who need additional insulin or who cannot tolerate IDegLira, insulin degludec will be used. Dose is titrated to achieve fasting normoglycemia.
  Arms: Intervention
Drug: Metformin — Dose is titrated to 2000 mg per day or maximal tolerated dose
  Arms: Intervention
Behavioral: Lifestyle Therapy — Lifestyle intervention includes individualized dietary and exercise advice targeting at least 5% weight loss with frequent visits and coaching for goal reinforcement, behavior modification and problem-solving
  Other Names: diet and exercise
  Arms: Intervention

SUMMARY:
The purpose of the study is to determine whether in patients with early type 2 diabetes, a short-term intensive metabolic intervention comprising IDegLira, metformin, and lifestyle approaches will be superior to standard diabetes therapy in achieving sustained diabetes remission.

DETAILED DESCRIPTION:
This is a multicentre, open-label, randomized controlled trial in 160 patients with recently-diagnosed T2DM. Participants will be randomized to 2 treatment groups: (a) a 16-week course of treatment with IDegLira, metformin and lifestyle therapy, and (b) standard diabetes therapy, and followed for a total of 68 weeks (1 year and 4 months). In all participants with HbA1C<7.3% at the 16 week visit, glucose-lowering medications will be discontinued and participants will be encouraged to continue with lifestyle modifications and regular glucose monitoring. Participants with HbA1C ≥ 7.3% at this visit or who experience hyperglycemia relapse after stopping drugs will receive standard glycemic management as informed by the current Canadian Diabetes Association clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. men and women aged 30-80 years;
2. T2D diagnosed within 5 years
3. stable T2D drug regimen in the 8 weeks before randomization;
4. HbA1c 6.5-9.5% on no glucose lowering drugs, or 6.5%-8.0% on up to 2 glucose lowering drugs;
5. body mass index ≥ 23 kg/m2;
6. ability and willingness to perform self-monitoring of capillary blood glucose (SMBG);
7. willingness to wear a continuous glucose monitor on at least 3 occasions;
8. ability and willingness to self-inject IDegLira and insulin;
9. provision of informed consent.

Exclusion Criteria:

1. current use of insulin therapy;
2. history of hypoglycemia unawareness, or severe hypoglycemia requiring assistance;
3. history of end-stage renal disease or eGFR<45 mL/min/1.73 m2 by MDRD formula;
4. active liver disease or elevated alanine transferase (ALT) levels ≥ 2.5 times the upper limit of normal at the time of enrolment;
5. history or clinical suspicion of pancreatitis or medullary thyroid cancer;
6. diagnosis or first degree relative with Multiple Endocrine Neoplasia Type 2 (MEN2);
7. history of diabetic retinopathy requiring photocoagulation, injection therapy or vitrectomy;
8. history of cardiovascular disease (unless cleared for a moderate intensity exercise program by a specialist) including: i. acute coronary syndrome, hospitalization for unstable angina, myocardial infarction, or revascularization with coronary artery bypass grafting or percutaneous coronary intervention; ii. peripheral vascular disease, valvular heart disease, cardiomyopathy, aortic dissection, tachyarrhythmias, bradyarrhythmias, prior stroke or TIA; iii. prior hospitalization for heart failure; or iv. ECG findings concerning for ischemic heart disease (i.e. pathological Q-waves, ST-segment-T-wave abnormalities in contiguous leads, left anterior hemiblock, left bundle branch block, second or third degree atrioventricular block).
9. history of any disease requiring frequent intermittent or continuous systemic glucocorticoid treatment;
10. history of bariatric surgery, or planned bariatric surgery in the next 1.5 years;
11. history of any major illness with a life expectancy of < 3 years;
12. history of injury or any other condition that significantly limits participant's ability to achieve moderate levels of physical activity;
13. excessive alcohol intake, acute or chronic;
14. currently pregnant, or breastfeeding, or not using a reliable method of birth control for the duration of the trial in all females with childbearing potential;
15. inability to take insulin degludec, liraglutide or metformin.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving drug-free diabetes remission | 28 weeks after randomization
  Drug-free diabetes remission is defined as HbA1C < 6.5 % off glucose-lowering agents for at least 12 weeks.

SECONDARY OUTCOMES:
Proportion of participants achieving drug-free diabetes remission | 28 weeks, 40 weeks, 52 weeks and 68 weeks after randomization
Proportion of participants achieving drug-free normoglycemia | 28 weeks, 40 weeks, 52 weeks and 68 weeks after randomization
  defined as HbA1C < 6.0% off glucose-lowering agents for at least 12 weeks.
Proportion of participants achieving drug-free diabetes regression | 28 weeks, 40 weeks, 52 weeks and 68 weeks after randomization
  defined as HbA1C <7.0% off glucose-lowering agents for at least 12 weeks.

OTHER OUTCOMES:
the time interval from randomization until any glucose lowering drug is restarted or relapse of hyperglycemia | Up to week 68
the time interval from the 16 week visit (i.e. when glucose lowering drugs are to be stopped) until any glucose lowering drug is restarted or relapse of hyperglycemia | Up to week 68
the change in HbA1c | 16, 28, 40, 52 and 68 week visit as well as the overall change
the change in weight | 16, 28, 40, 52 and 68 week visit as well as the overall change
the change in waist circumference | 16, 28, 40, 52 and 68 week visit as well as the overall change
the change in hip circumference | 16, 28, 40, 52 and 68 week visit as well as the overall change
the change in body mass index | 16, 28, 40, 52 and 68 week visit as well as the overall change
the change in coefficient of variation over 2 weeks (defined as 4-8 mmol/l), based on up to 2 weeks of Abbott Freestyle Libre ProTM sensor wear | from randomization until the 6, 16, 28 and 52 week visit
the change in interquartile range over 2 weeks (defined as 4-8 mmol/l), based on up to 2 weeks of Abbott Freestyle Libre ProTM sensor wear | from randomization until the 6, 16, 28 and 52 week visit
the change in time range over 2 weeks (defined as 4-8 mmol/l), based on up to 2 weeks of Abbott Freestyle Libre ProTM sensor wear | from randomization until the 6, 16, 28 and 52 week visit

CONTACTS AND LOCATIONS:
Overall Officials: Zubin Punthakee, MD, Principal Investigator — McMaster University; Hertzel Gerstein, MD, Study Chair — McMaster University
Locations (8):
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - St. Joseph's Hospital, London, Ontario
  - Western University, London, Ontario
  - LMC Manna Research, Oakville, Ontario
  - The Ottawa Hospital, Ottawa, Ontario